CLINICAL TRIAL: NCT02457741
Title: A Simple Approach to Estimate Alveolar Recruitability in Patients With Acute Respiratory Distress Syndrome: a Validation Study
Brief Title: Validation of a Simple Approach to Estimate Alveolar Recruitability in ARDS Patients
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: REB# 15-074
Record Dates: First submitted 2015-05-19; First posted 2015-05-29 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Mechanical ventilation; PEEP; Respiratory mechanics; End-expiratory lung volume
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will test the validity of a new approach to assess alveolar recruitability at the bedside in comparison to direct measurements of lung volume and derecruitment.

DETAILED DESCRIPTION:
Background: Acute respiratory distress syndrome (ARDS) is characterized by a major loss of lung volume due to alveolar flooding, atelectasis and consolidation[1]. Positive end-expiratory pressure (PEEP) is applied to recruit non-aerated or poorly aerated lung tissue, and thus may improve gas exchange in patients with ARDS[2]. However, PEEP may also be harmful by overdistending the previously open lung tissue. The potential effectiveness and benefit of high PEEP levels depends on the patient's recruitability. Previous techniques for assessing recruitability are usually reserved for clinical research (computed tomography, multiple pressure-volume curves)[3-4] or need special equipment. A simple, feasible bedside method to assess the individual needs for PEEP in terms of recruitability seem essential to improve the prognosis of this syndrome. The investigators therefore propose a simplified approach derived from our previous study[5] to estimate alveolar recruitability at the bedside.

Objectives: The major aim is to test the hypothesis that this simplified approach is a valid method for assessing alveolar derecruitment at the bedside in comparison to direct measurements of lung volume and derecruitment.

Methods: This physiological study will enroll 30 patients from the three Intensive Care Units at St. Michael's Hospital in two years. All patients will be passively ventilated at two PEEP levels (15 cmH2O and 5 cmH2O) and the plateau pressure will be limited to less than 35 cmH2O. Respiratory mechanics, lung volumes (using the nitrogen washout/washin technique), quasi-static Pressure-Volume curves, lung ultrasound, and arterial blood gases will be assessed at each PEEP level. In patients who already have an esophageal catheter in place, Pes will also be measured.

Data Analysis: The primary endpoint is the correlation and bias between the Vder estimated by our approach and the one measured by the multiple P-V curves technique through paired tests, correlations and Bland and Altman analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients > 16 years of age
* Moderate-to-severe ARDS as per the Berlin definition (Partial pressure of oxygen (PaO2)/Fraction of inspired oxygen (FiO2) < 200 mmHg) and within 10 days of onset
* Receiving assist/control mechanical ventilation (volume or pressure) with continuous sedation and an established arterial line

Exclusion Criteria:

* Pneumothorax with fistula or likely to require a chest tube
* Severe hemodynamic instability (> 30% increase in vasopressors in the last 6 hours or norepinephrine > 0.5 µg/kg/min)
* PaO2/FiO2 < 80 mmHg
* Severe or very severe Chronic Obstructive Pulmonary Disease according to the GOLD criteria (stage III: Forced expiratory volume at one second (FEV1) 30-50% predicted; stage IV: FEV1 < 30% predicted)
* Known or highly suspected elevated intracranial pressure (> 18 mmHg)

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Moderate-to-severe ARDS patients as per the Berlin definition
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The derecruited volume estimated (Vder,est) by our new approach will be compared with the one measured by the multiple P-V curves technique (Vder,meas) | 90-120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brochard, MD, Principal Investigator — Unity Health Toronto
Locations (3):
- St. Michael's Hospital, Toronto, Ontario, Canada
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China
- Centre Hospitalier Universitaire - CHU Angers, Angers, France

REFERENCES:
- [Background] Chen L, Brochard L. Lung volume assessment in acute respiratory distress syndrome. Curr Opin Crit Care. 2015 Jun;21(3):259-64. doi: 10.1097/MCC.0000000000000193. PMID 25827584
- [Background] Ashbaugh DG, Bigelow DB, Petty TL, Levine BE. Acute respiratory distress in adults. Lancet. 1967 Aug 12;2(7511):319-23. doi: 10.1016/s0140-6736(67)90168-7. No abstract available. PMID 4143721
- [Background] Gattinoni L, Caironi P, Cressoni M, Chiumello D, Ranieri VM, Quintel M, Russo S, Patroniti N, Cornejo R, Bugedo G. Lung recruitment in patients with the acute respiratory distress syndrome. N Engl J Med. 2006 Apr 27;354(17):1775-86. doi: 10.1056/NEJMoa052052. PMID 16641394
- [Background] Maggiore SM, Jonson B, Richard JC, Jaber S, Lemaire F, Brochard L. Alveolar derecruitment at decremental positive end-expiratory pressure levels in acute lung injury: comparison with the lower inflection point, oxygenation, and compliance. Am J Respir Crit Care Med. 2001 Sep 1;164(5):795-801. doi: 10.1164/ajrccm.164.5.2006071. PMID 11549535
- [Background] Dellamonica J, Lerolle N, Sargentini C, Beduneau G, Di Marco F, Mercat A, Richard JC, Diehl JL, Mancebo J, Rouby JJ, Lu Q, Bernardin G, Brochard L. PEEP-induced changes in lung volume in acute respiratory distress syndrome. Two methods to estimate alveolar recruitment. Intensive Care Med. 2011 Oct;37(10):1595-604. doi: 10.1007/s00134-011-2333-y. Epub 2011 Aug 25. PMID 21866369
- [Derived] Chen L, Del Sorbo L, Grieco DL, Junhasavasdikul D, Rittayamai N, Soliman I, Sklar MC, Rauseo M, Ferguson ND, Fan E, Richard JM, Brochard L. Potential for Lung Recruitment Estimated by the Recruitment-to-Inflation Ratio in Acute Respiratory Distress Syndrome. A Clinical Trial. Am J Respir Crit Care Med. 2020 Jan 15;201(2):178-187. doi: 10.1164/rccm.201902-0334OC. PMID 31577153